CLINICAL TRIAL: NCT03324412
Title: A 24-Week, Multicenter ,Double Blind, Randomized Study to Determine the Effects and Security of TwHF and MTX Treating Rheumatoid Arthritis
Brief Title: Efficacy and Safety of TwHF and MTX in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, director, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z161100000516020-2
Record Dates: First submitted 2017-10-25; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of MTX (Active Comparator): Patients were treated with methotrexate (MTX)and Tripterygium wilfordii Hook F（TwHF）placebo.
  Interventions: Drug: Treatment of MTX
- Treatment of MTX and TwHF (Experimental): Patients were treated with methotrexate (MTX)and Tripterygium wilfordii Hook F（TwHF).
  Interventions: Drug: Treatment of MTX and TwHF

INTERVENTIONS:
Drug: Treatment of MTX — Methotrexate: 10-15mg per week according to patient's weight, oral, for 24 weeks.Tripterygium wilfordii Hook F（TwHF）placebo：20mg， 3 times a day, oral, for 24 weeks.
  Arms: Treatment of MTX
Drug: Treatment of MTX and TwHF — Methotrexate : 10-15mg per week according to patient's weight, oral, for 24 weeks.Tripterygium wilfordii Hook F（TwHF）：20mg， 3 times a day, oral, for 24 weeks.
  Arms: Treatment of MTX and TwHF

SUMMARY:
Rheumatoid Arthritis (RA) is an autoimmune disease that results in a chronic inflammatory disorder that may affect many synovial joints, and may cause serious disability. It has been confirmed that Tripterygium Wilfordii has effects of anti-inflammatory, immunosuppressive and cartilage protection. This is a multicenter ,double Blind, randomized study to evaluated the efficacy and safety of Tripterygium Wilfordii in treating of patients with rheumatoid arthritis (RA) and establish a prediction model for Tripterygium Wilfordii response of rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Two arms were included in this study. Active Comparator: treatment of MTX Patients were treated with methotrexate (MTX)and Tripterygium wilfordii Hook F（TwHF）placebo.Experimental: treatment of TwHF Patients were treated with methotrexate (MTX) and Tripterygium wilfordii Hook F（TwHF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis as determined by the 1987 or 2010 ACR classification criteria;
* No male or female fertility requirements, or around menopause women;
* Patients with mild-to-moderate activity, 2.6 < DAS28≤5.1;
* No serious system involved, such as severe pericardial effusion, interstitial lung disease, renal tubular acidosis, atrophic gastritis, autoimmune liver disease, etc;
* Within a month before the selected participants did not attend any drugs

Exclusion Criteria:

* Patients with cancer or other malignant disease such as cardiovascular, hematopoietic, liver and kidney disease, and psychopath
* Active or chronic infection, including HIV, hepatitis C virus, hepatitis B virus, tuberculosis
* Previous treated with tripterygii, glucocorticoid or biologic disease-modifying antirheumatic drug (DMARD) in 3 months.
* Previous treated with Tripterygium Wilfordii or MTX
* Patients with retinopathy.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2017-10-28 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
The change from Baseline to week 24 in Disease Activity Score (DAS28) | 0 weeks, 4 weeks，12 weeks, 24 weeks,52 weeks
  Disease Activity Score for 28-joint counts was based on the erythrocyte sedimentation rate(ESR) (DAS28-4[ESR])

SECONDARY OUTCOMES:
The proportion of patients achieving ACR20/50/70 | 0 weeks, 4 weeks，12 weeks, 24 weeks
  ACR20/50/70 is referred to American College of Rheumatology Criteria
The change in Health Assessment Questionnaire (HAQ) score | 0 weeks, 4 weeks，12 weeks, 24 weeks,52 weeks
  HAQ scores ranges from 0 to 3, with higher scores indicating greater disability
The change in Sharp score | 0 week,24 weeks,52 weeks
  The change in X-Ray from baseline to week 24 and 52.
The number of adverse events | 24 weeks
  The number of adverse events that are related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No